CLINICAL TRIAL: NCT01743079
Title: The Efficacy and Safety of Telbivudine and Lamivudine Use in Highly Viremic Mothers to Prevent Hepatitis B Transmission
Brief Title: Study of Telbivudine and Lamivudine to Prevent Vertical Transmission of Hepatitis B
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Beijing YouAn Hospital (Other)
Collaborators: New Discovery LLC (Industry)
Responsible Party: Principal Investigator, Hua Zhang, Professor, Beijing YouAn Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20080810
Record Dates: First submitted 2012-12-03; First posted 2012-12-06 (Estimated); Last update posted 2013-07-30 (Estimated); Status verified 2013-07

CONDITIONS: Chronic Hepatitis B; Late Pregnancy; Transmission; Complication
Keywords: Telbivudine; Lamivudine; safety; efficacy; pregnancy
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — Telbivudine; Lamivudine; lipoarabinomannan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Telbivudine (Experimental): Mother receives telbivudine 600mg per day. Infant receives standard immunoprophylaxis
  Interventions: Drug: Telbivudine
- Lamivudine (Experimental): Mother receives lamivudine 100mg per day. Infant receives standard immunoprophylaxis.
  Interventions: Drug: Lamivudine
- No antiviral treatment (No Intervention): Mother receives no antiviral treatment. Infant receives standard immunoprophylaxis

INTERVENTIONS:
Drug: Telbivudine — LdT 600mg QD
  Other Names: LdT
  Arms: Telbivudine
Drug: Lamivudine — LAM 100mg QD
  Other Names: LAM
  Arms: Lamivudine

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of telbivudine and lamivudine use during late pregnancy for the prevention of HBV perinatal transmission in highly viraemic mothers.

DETAILED DESCRIPTION:
This study enrolls HBV mono-infected pregnant women cohorts managed in outpatient clinics/delivery unit at YouAn Hospital in Beijing. Subjects are prospectively followed from gestation week 26 to postpartum week 52. Treatment naïve mothers with HBV DNA > 6 log10 c/mL and normal ALT are eligible. Mothers with abnormal fetus, cirrhosis or evidence of hepatocellular carcinoma (HCC) are excluded. At gestation week 28, mothers will receive telbivudine (LdT) 600 mg per day or lamivudine (Lam) 100 mg per day until postpartum 4 or no treatment as per their preference. All infants will receive standard immunoprophylaxis. Data is collected from patient records using data extraction forms. Primary endpoints are vertical transmission rates at infants' age of 52 week and the safety of telbivudine or lamivudine use.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 20-40 years old
2. HBsAg, HBeAg positive and HBV DNA >6 log10 copies/ml
3. Gestational age: 26-28 weeks with normal fetus
4. Willing to consent for the study

Exclusion Criteria:

1. Elevated ALT
2. Antiviral treatment experience patients
3. Co-infection with HAV, HCV,HDV, HIV
4. Concurrent treatment with immune modulators, cytotoxic drugs, or steroids
5. Clinical signs of threatened miscarriage in early pregnancy
6. Clinical evidence of cirrhosis and/or hepatocellular carcinoma

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 700 (Actual)
Dates: Start 2009-01; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Safety on fetal exposure of telbivudine and lamivudine and vertical transmission rate from mother to child | From gestation week 26 to postpartum week 52

SECONDARY OUTCOMES:
percentage of mothers with serum HBV DNA level reduction, ALT within normal range and HBeAg and/or HBsAg negativity with or without seroconversion | From gestation week 26 to pastpartume week 52

CONTACTS AND LOCATIONS:
Overall Officials: Calvin Pan, MD, Study Director — Division of Liver Diseases, Mount Sinai School of Medicine, Flushing, NY; Hua Zhang, MD, Principal Investigator — Beijing YouAn Hospital
Locations (1):
- Beijing YouAn Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Zhang H, Pan CQ, Pang Q, Tian R, Yan M, Liu X. Telbivudine or lamivudine use in late pregnancy safely reduces perinatal transmission of hepatitis B virus in real-life practice. Hepatology. 2014 Aug;60(2):468-76. doi: 10.1002/hep.27034. Epub 2014 Jan 27. PMID 25187919